CLINICAL TRIAL: NCT00612833
Title: A Randomized Controlled Trial of Three Vasectomy Techniques
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: FHI 360 participation in the study was terminated due to lack of funding
Sponsor: FHI 360 (Other)
Collaborators: Indian Council of Medical Research (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: FHI-9980
Record Dates: First submitted 2008-01-29; First posted 2008-02-12 (Estimated); Last update posted 2013-09-10 (Estimated); Status verified 2013-09

CONDITIONS: Contraception
Keywords: Vasectomy; Male contraception; Contraceptive effectiveness; Semen analysis; Surgical techniques; Fascial interposition; Cautery; The relative contraceptive effectiveness of three methods of occluding the vas, in the context of a no-scalpel vasectomy procedure.

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- cautery excision with fascial interposition (Active Comparator): Contraception using cautery and excision with fascial interposition
  Interventions: Procedure: Vasectomy occlusion techniques
- B (Active Comparator): Cautery and excision without fascial interposition
  Interventions: Procedure: Vasectomy occlusion techniques
- C (Active Comparator): Ligation and excision with fascial interposition
  Interventions: Procedure: Vasectomy occlusion techniques

INTERVENTIONS:
Procedure: Vasectomy occlusion techniques — Cautery and excision with fascial interposition Cautery and excision without fascial interposition Ligation and excision with fascial interposition

SUMMARY:
This study will be a randomized, controlled multicenter trial, conducted jointly by the Indian Council of Medical Research, New Delhi and Family Health International, which will compare three vasectomy occlusion techniques, all using the no-scalpel vasectomy (NSV) approach to isolation of the vas:

1. ligation and excision of about 1 cm of the vas, with fascial interposition;
2. intraluminal thermal cautery with excision of about 1 cm of the vas;
3. intraluminal thermal cautery with excision of about 1 cm of the vas combined with fascial interposition.

A total of 1500 healthy, sexually active men at least 21 years old who have chosen vasectomy as a means of contraception will be recruited at four to six study sites in India. The success of the vasectomy procedure will be determined based on semen analysis results. All men should have semen analyses at 8 and 12 weeks post-vasectomy. All men will be asked to attend a final visit at 12 months.

DETAILED DESCRIPTION:
This study will be a randomized, controlled multicenter trial, conducted jointly by the Indian Council of Medical Research, New Delhi and Family Health International, which will compare three vasectomy occlusion techniques, all using the no-scalpel vasectomy (NSV) approach to isolation of the vas:

1. ligation and excision of about 1 cm of the vas, with fascial interposition;
2. intraluminal thermal cautery with excision of about 1 cm of the vas; and,
3. intraluminal thermal cautery with excision of about 1 cm of the vas combined with fascial interposition.

A total of 1500 healthy, sexually active men at least 21 years old who have chosen vasectomy as a means of contraception will be recruited at four to six study sites in India. The success of the vasectomy procedure will be determined based on semen analysis results. All men should have semen analyses at 8 and 12 weeks post-vasectomy. All men will be asked to attend a final visit at 12 months.

ELIGIBILITY:
Inclusion Criteria:

1. Freely consent to participate in the study and sign an informed consent form
2. Be at least 21 years old
3. The couple should have at least one living child greater than one year of age
4. With his partner be willing to use an alternate method of contraception until success is confirmed
5. Be willing to return for follow-up visits at 1, 8, 12 and 52 weeks post-vasectomy, and at 16, 20 and 24 weeks if needed
6. Be willing to submit semen samples collected by masturbation in the clinic according to the study follow-up schedule
7. Be able to understand the procedures and study requirements

Exclusion Criteria:

1. Has a condition that in the opinion of the investigator permanently or temporarily contraindicates participation in the study, e.g., depression or poorly-controlled diabetes
2. History of surgery involving the vas or testes (including previous vasectomy)
3. Previous injury or significant abnormality of the scrotum
4. Clinical evidence of an acute sexually transmitted infection; however a man may be admitted to the study after resolution of the acute condition.
5. Local genital infections such as balanitis, scrotal skin infection, epididymitis, or orchitis, but a man may be admitted after resolution of an acute infection
6. History of coagulation or other bleeding disorders
7. Large varicocele, hydrocele, filariasis or elephantiasis of scrotum, or intrascrotal mass
8. Acute systemic infection (including gastroenteritis), but a man may be admitted after resolution of the condition
9. Currently taking or planning to take any type of systemic medication which could affect sperm count (e.g. anabolic steroids)

Min Age: 21 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2009-01

PRIMARY OUTCOMES:
Sperm concentration in semen | 12 weeks

SECONDARY OUTCOMES:
Safety | up to 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Chander Shekhar, MD, Principal Investigator — ICMR; David C. Sokal, MD, Principal Investigator — FHI 360
Locations (5):
- India (5):
  - Post Graduate Institute of Medical Sciences, Rohtak, Haryana
  - Maulana Azad Medical College, New Delhi, National Capital Territory of Delhi
  - St. Stephens Hospital, New Delhi, National Capital Territory of Delhi
  - Civil Hospital,, Amritsar, Punjab
  - E. S.T.N.M. Hospital, Gangtok, Gangtok, Sikkim

REFERENCES:
- See also: Related Info — http://www.fhi.org